CLINICAL TRIAL: NCT03602209
Title: Short vs. Long Antibiotic Treatment of Implant-free Osteoarticular Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Ilker Uckay, Attending, Docent Dr. med. Ilker Uçkay, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. 14-198
Record Dates: First submitted 2017-01-17; First posted 2018-07-26 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Implant Infection
Keywords: implant-related infections; orthopaedics; implant removal; antibiotic duration; outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 weeks of treatment (Experimental)
  Interventions: Procedure: Removal of infected implant; Drug: Antibiotic durations
- 6 weeks of treatment (Active Comparator)
  Interventions: Procedure: Removal of infected implant; Drug: Antibiotic durations

INTERVENTIONS:
Procedure: Removal of infected implant
Drug: Antibiotic durations

SUMMARY:
The investigators tested the working hypothesis if 4 weeks of systemic antibiotic treatment in implant-related orthopaedic infections is non-inferior to 6 weeks after complete removal of the infected implant. Randomization 1:1.

The study is completed. It halted prematurely and will not resume; participants are no longer being examined or receiving intervention.

DETAILED DESCRIPTION:
Former description of the study (now completed)

Osteoarticular infections related to orthopaedic implants are associated with substantial morbidity, prolongation of hospital stay, and additional costs. Due to the increasing number of patients with orthopaedic implants in Switzerland, similar to the rest of Europe and elsewhere, the number of infections is expected to increase. While the surgical treatment of these infections has been well studied, the ideal duration of antibiotic therapy after removal (explantation) of the infected implant remains unknown. For almost 40 years, the recommended total duration of post-explantation antibiotic therapy has been 6 weeks. This recommendation is based on expert's personal experience rather than on prospective randomized studies. Shorter treatment would decrease antibiotic-related adverse events and costs hospital stay for patients awaiting an eventual reinsertion of a new implant. If physicians and surgeon prescribe antibiotics for 6 weeks, this duration should be at least supported by evidence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥17 years old)
* Total removal of the implant

Exclusion Criteria:

* Primary native joint septic arthritis;
* Co-trimoxazole prophylaxis because of immunosuppression;
* Left-side endocarditis;
* Persistent implant material in the infected area.
* Infections with tuberculosis; mycobacteria; fungi; brucellosis; borreliosis; nocardiosis; and mycoplasmal osteosynthesis infections

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Remission of infection | 12 months
  Clinical evaluation
Adverse events | 12 months
  Clinical adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mayahi M, Betz M, Muller DA, Stern R, Tahintzi P, Bernard L, Hoffmeyer P, Suva D, Uckay I. Remission rate of implant-related infections following revision surgery after fractures. Int Orthop. 2013 Nov;37(11):2253-8. doi: 10.1007/s00264-013-2092-1. Epub 2013 Sep 20. PMID 24052163